CLINICAL TRIAL: NCT06964594
Title: A Randomized Controlled Trial Study Comparing Adnexal Surgery by vNOTES or Laparoscopy
Acronym: ADNOLA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Andrea Stuart, Associate Professor, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-00965-01
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Cysts; Laparoscopic Gynecologic Surgery; vNOTES
Keywords: ADNOLA - A randomized controlled trial study comparing adnexal surgery by vNOTES or laparoscopy
MeSH Terms: conditions — Ovarian Cysts

STUDY DESIGN:
Intervention Model Description: Pragmatic multicentre two-armed superiority randomized controlled trail. No blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic Adnexal surgery (Active Comparator)
  Interventions: Procedure: vNOTES adnexal surgery

INTERVENTIONS:
Procedure: vNOTES adnexal surgery — New minimalinvasive technique

SUMMARY:
The aim with the study is to compare postoperative pain after vNOTES adnexal surgery versus laparoscopic adnexal surgery.

Women aged 18 and above with an indication for adnexal surgery for benign gynecological pathology or prophylactic reasons will be able to participate.

After surgery the participants will answer a questioner, twice a day in seven days, about postoperative pain and how many units of analgesics they used.

Adnexal surgery is one of the most common surgical procedures performed in women and can either be performed to treat pathology as ovarian cysts or prophylactically in case of hereditary genetic alterations.

A laparoscopic technique is currently considered as gold standard for adnexal procedures. The latest advancement in minimally invasive surgery is vNOTES (vaginal natural orifice transluminal endoscopy), in which the entrance to the abdomen is performed by an anterior or more commonly posterior colpotomy rather than via the abdominal wall. The NOTABLE trial was a RCT showing that vNOTES adnexectomy was non-inferior to laparoscopy for successful removal of benign adnexa without conversion (Baekelandt). vNOTES adnexectomy had shorter surgical time, less use of analgesics and lower self-assessed VAS scores the first week post-operatively. The aim with our study is to compare postoperative pain after vNOTES versus laparoscopic adnexal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Female aged 18 years or above.
* Diagnosed with adnexal pathology or subject for prophylactic BSO.

Exclusion Criteria:

* Female participant who is pregnant or planning pregnancy during course of the trial.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Patients taking opioids or other painkillers routinely pre-operatively.
* Patients with chronic pelvic pain.
* Patients with surgical contraindication; previous hysterectomy, history of rectal surgery, suspected or confirmed endometriosis, suspected malignancy, suspected obliteration of the pouch of Douglas following severe PID or other causes, active lower genital tract infection, pregnancy.
* Failure to provide written informed consent prior to surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Pain postoperatively by a VAS-scale | 7 days postoperative
  To compare postoperative pain after adnexal surgery performed by vNOTES or laparoscopy

SECONDARY OUTCOMES:
Painkillers used (amount) | 7 days postoperatively
  Units of non-opioid analgesics Units of postoperative opioids
Perioperatively complications | Perioperatively
  The incidence of intra-operative complications, i.e. any adverse event before the end of the surgical intervention including injury to the bladder, ureter, bowel, or intrapelvic/intra-abdominal vessels, as a dichotomous outcome.
Operation time | Perioperatively
  Operation time, measured as the time in minutes from the insertion of the bladder catheter to the end of vaginal/abdominal wound closure, as a continuous outcome.
Postoperative complications | 6 weeks postoperatively
  Postoperative complications: major bleeding or pelvic hematoma requiring transfusion. Infections of the vaginal incision, abdominal wall or wound, urinary tract, chest, or febrile episodes/unspecified infections. Thromboembolism. Postoperative ileus or wound dehiscence. Classified according to the Clavien- Dindo, classification as a dichotomous outcome.
Readmission | 6 weeks after surgery
  The rates of readmission requiring hospitalization for at least 24 hours for any adverse event causally related to the gynaecological intervention during the first six weeks after surgery, as a dichotomous outcome.
Conversion rate | Perioperatively
  Conversion rates: the proportion of women treated by any other approach than the allocated technique as randomized, as a dichotomous outcome. vNOTES will most likely be converted to LSC and LSC to open surgery
Surgeon's experience | Perioperatively
  Surgeon's experience of comfort and flow measured by a 0 to 10 mm VAS scale

IPD SHARING:
Plan to Share IPD: No